CLINICAL TRIAL: NCT07352397
Title: The Effect of Inhaled Lavender Oil, Rosemary Oil, and Their Combination in Reducing Dental Anxiety and Pain in Pediatric Dental Patients (A Randomized Controlled Clinical Trial)
Brief Title: Inhaled Lavender Oil, Rosemary Oil, and Their Combination in Reducing Dental Anxiety and Pain in Pediatric Dental Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1188-11/2025
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Experimental)
  Interventions: Other: Lavender group
- Group II (Experimental)
  Interventions: Other: Rosemary group
- Group III (Experimental)
  Interventions: Other: Combination of both lavender and rosemary
- Group IV (Active Comparator)
  Interventions: Other: No essential oils

INTERVENTIONS:
Other: Lavender group — Children in this group will be inhaled 0.5 ml of prepared mixture (of Lavandula Angustifolia+ Sweet Almond carrier oil ) on a cotton pad attached to the facial steamer .
  Arms: Group I
Other: Rosemary group — Children in this group will be inhaled 0.5 ml of prepared mixture (of Rosmarinus Officinalis + Sweet Almond carrier oil ) on a cotton pad attached to the facial steamer
  Arms: Group II
Other: Combination of both lavender and rosemary — Children in this group would be inhaled 0.5 ml of prepared mixture (of Lavandula Angustifolia and Rosmarinus Officinalis + Sweet Almond carrier oil) on a cotton pad attached to the facial steamer .
  Arms: Group III
Other: No essential oils — Children in this group will be inhaled 0.5 mL of the carrier oil (Sweet Almond ) on a cotton pad attached to the facial steamer .
  Arms: Group IV

SUMMARY:
Background: Dental anxiety and pain are common concerns in pediatric dentistry. These issues can lead to negative experiences for children and can make it difficult for them to cooperate during treatment. While medications can help manage these symptoms, it can also have side effects. This highlights the need for safe and effective complementary treatments. Aromatherapy, particularly with lavender and rosemary oils, has demonstrated anxiolytic and analgesic properties in different fields. However, their effect in helping children cope with dental anxiety and pain during procedures requiring local anesthesia has not yet been thoroughly studied.

Purpose: This study aims to investigate the efficacy of inhaled lavender oil, rosemary oil, and their combination in reducing dental anxiety and pain in children receiving local anesthesia for extraction of lower primary molar

ELIGIBILITY:
Inclusion Criteria:

* Frankl behavioural rating score 2 or 3 during preoperative assessment.
* Healthy children ASAI.
* Children without a previous dental history.
* Children presenting with at least one mandibular molar indicated for extraction. (43)
* Completion of the written informed consent form by parents/guardian.

Exclusion Criteria:

* Children with colds, asthma, and any other respiratory diseases.
* Children who took NSAIDs or analgesic drugs in the last 8 hours before treatment.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety scores | up to 1 week
  Venham scale will be used. it ranges from 0 (relaxed) to 5 (Child out of contact with the relaity of threat)

SECONDARY OUTCOMES:
Change in anxiety scores (by children) | up to 1 week
  Comprises a row of five faces ranging from very happy (score 1) to very unhappy (score 5)
Change in pain scores | up to 1 week
  FLACC scale. It is an objectively pain assessment Scale .The scale quantifies pain by observing five distinct behavioral categories: face, legs, activity, cry, and consolability. Each category is assigned a score from 0 to 2, which are then summed to yield a total pain score ranging from 0 to 10.
Change in heart rate | During procedure
  it will be used by pulse oximeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt